CLINICAL TRIAL: NCT06487130
Title: Virtual perI-/Menopause Registry of AusTrALia
Acronym: VITAL
Status: Recruiting | Type: Observational
Sponsor: Bespoke Clinical Research (Industry)
Responsible Party: Principal Investigator, Erin Morton, Associate Professor, Bespoke Clinical Research
Other Study IDs: VITAL-Oz
Record Dates: First submitted 2023-08-14; First posted 2024-07-05 (Actual); Last update posted 2024-07-05 (Actual); Status verified 2024-07

CONDITIONS: Menopause; Perimenopausal Disorder; Postmenopausal Symptoms; Health Knowledge, Attitudes, Practice; Healthy Aging; Health Care Utilization; Health Care Seeking Behavior; Mental Health Impairment; Mental Deterioration; Mental Health Issue; Osteoporosis, Postmenopausal; Diabetes Mellitus Risk; Diabetes Mellitus, Type 2; Dementia; Cardiovascular Diseases; Menopause Related Conditions; Hot Flashes; Hot Flushes Aggravated; Economic Burden; Social Stigma
MeSH Terms: conditions — Behavior; Patient Acceptance of Health Care; Cognitive Dysfunction; Osteoporosis, Postmenopausal; Diabetes Mellitus, Type 2; Dementia; Cardiovascular Diseases; Hot Flashes; Financial Stress; Social Stigma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 50 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Menopause/Post-menopause: Menopause/Post-menopause, born with ovaries
  Interventions: Other: N/A Observational Registry
- Peri-menopause: Peri-menopause, born with ovaries
  Interventions: Other: N/A Observational Registry
- Pre-menopause: Pre-menopause, born with ovaries
  Interventions: Other: N/A Observational Registry
- Other: Not born with ovaries
  Interventions: Other: N/A Observational Registry

INTERVENTIONS:
Other: N/A Observational Registry — Registry participants may select to be contacted for future research and/or embedded clinical trials. Such interventions will require associated ethics review & approval.

SUMMARY:
13 million (50.7%) Australians are born with ovaries, 14% (~3 million) are currently aged 40-59 yrs, & all such who live to midlife will experience menopause, defined as >12 months without a period. Peri-menopause (peri), typically occurs 5 yrs before menopause as hormone levels decrease. As with oestrogen, peri symptoms can affect every bodily system; e.g. depression/anxiety, diminished mental function, irregular periods, hot flushes, sleep problems, vaginal atrophy & urinary urgency. These symptoms are linked with lower quality of life & significantly higher work impairment; a third experiencing symptoms so severe as to impede daily life & increase risk of suicide. Lifetime increased risks of diabetes, heart disease, osteoporosis & dementia are also associated with menopause, yet it remains disconcertingly poorly studied.

The investigators propose to create a world-first, cutting-edge, consumer-driven, Virtual peri-/menopause registry of AusTrALia (VITAL). The unique design will enable consumers to determine VITAL's questions, encourage secure revelation of private data e.g. vaginal & mental health symptoms, & to direct priorities for research, education, & health service improvements. VITAL will thus deliver optimal assessments of incidence, prevalence & impact.

The participating consumers, researchers, clinical specialists, policy makers, & modern virtual data infrastructure enable this unique & innovative registry design, future translation to improved community health, & promote awareness & collaborative synergies. Leveraging the investigators' critical range of expertise & ongoing feedback opportunities for both participants & stakeholder partnerships, the investigators will create a ground-breaking platform that:

* empowers the consumer voice and priorities,
* enables peri-/menopause research to extend beyond existing niche focuses,
* evidences the true impact of peri-/menopause across the nation,
* evolves healthcare services and outcomes, &
* educates community, clinicians, & policy-makers. After Australian registry establishment, the investigators will expand VITAL to mirror it in other nations while still protecting individual's data the right way, but so all can learn & apply the best aspects of care from across the world.

DETAILED DESCRIPTION:
In the Virtual Peri-Menopause Registry of Australia -VITAL- the investigators will:

1. Co-create an innovative, multidisciplinary, ongoing digital epidemiological platform & repository of Australian peri-/menopausal health, centred on relevance to the community;
2. Establish incidence, prevalence & impact of Australian peri-/menopause symptomology, associated disease risk factors, & healthcare system pathways, via secure participant input, encouraging safe revelation of personal data, e.g. symptoms, impairment, substandard care;
3. Determine & define community consensus priorities in related healthcare & associated policy.
4. Disseminate not only results, but ensure accessibility of the data from the national registry to authorised, relevant & ethical investigations to streamline research & in turn, translate to community healthcare outcomes, e.g. community education, clinical advice, policies, data linkage with significant datasets and/or registries e.g. cardiac, cancer, ageing, Medicare etc.

ELIGIBILITY:
Inclusion Criteria:

* Any Australian over 18 years of age.

Exclusion Criteria:

* None.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Although most questions are targeted towards those in peri-/menopause, other members from the community, clinical, research, employment or other areas can also provide valuable input through participative responses to a smaller number of questions.
  Note "Australian" includes Australian residents utilising the Australian healthcare system.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2023-08-03 (Actual); Primary Completion 2073-08 (Estimated); Study Completion 2073-08 (Estimated)

PRIMARY OUTCOMES:
Australian peri-/menopause experience as measured by qualitative self-report generated via participation & feedback of a critical mass of at least 10,000 registry participants, broadly representative of the Australian population. | Through input completion per participant, an average of 4 years
  Determination of the Australian peri-/menopause experience.

SECONDARY OUTCOMES:
Registry feasibility as measured by numbers of registry entries. | Through study completion, ongoing at least quarterly for a minimum of 10 years post-registry commencement.
  Registry feasibility shown by increasing Australian participation

CONTACTS AND LOCATIONS:
Overall Officials: Erin B Morton, PhD,Medicine, Study Director — Bespoke Clinical Research
Locations (1):
- Bespoke Clinical Research. Community-driven from every Australian across the country. Registry led from Adelaide, Adelaide, Australia

IPD SHARING:
Plan to Share IPD: Yes
Individual Participant Data collected during the trial may be shared but only if that individual participant specifically consented to it, & only after approval decisions from both Ethics Committee & VITAL Steering Committee review. Otherwise any sharing and/or publication of this data will be deidentified and/or aggregated as appropriate.
Time Frame: Start dates: As appropriate to minimum data level reached for the question of interest.
  End dates: At end of registry unless particular parameters are removed via amendment during annual conduct, whereupon 15 years after final collection.
Access Criteria: Detailed requests must be submitted with ethics approval to the VITAL Steering Committee for review consideration. Sharing will be on hold by default until otherwise specified in VITAL information including public-facing webpage. Only IPD with individual-level consent will be shared. Otherwise any sharing and/or publication of VITAL data will be deidentified and/or aggregated as appropriate. Upon reaching internally-defined minimum data levels, more information on the IPD sharing request processes will be made available on the VITAL website.
URL: https://bespokeclinicalresearch.com.au/vitalimpact/

REFERENCES:
- See also: VITAL Research: co-creating healthcare improvement. — https://bespokeclinicalresearch.com.au/vitalimpact/